CLINICAL TRIAL: NCT07305922
Title: Delayed Cerebral Infarction Beyond Endoluminal Spasmolysis and Induced Hypertension
Acronym: Decibel
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Rudberg, Senior Consultant, Research Group Leader, Karolinska Institutet
Other Study IDs: 2025-4055
Record Dates: First submitted 2025-12-07; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Aneurysm Hemorrhage; Cerebral Vasospasm After Subarachnoid Hemorrhage
Keywords: Transcranial Doppler; Endoluminal Spasmolysis; Induced Hypertension; Multimodal Neuromonitoring
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with emerging or established severe cerebral vasospasm after subarachnoid haemorrhage
  Interventions: Drug: Induced hypertension with norepinephrine; Drug: Endoluminal Spasmolysis

INTERVENTIONS:
Drug: Induced hypertension with norepinephrine — Induced hypertension with norepinephrine and/or dobutamine to attain clinically established goals of cerebral perfusion pressure in a stepwise fashion, according to clinical routine.
Drug: Endoluminal Spasmolysis — Endoluminal spasmolysis of cerebral arteries using i.a. Nimodipine, according to clinical protocol and neurointerventionist discretion.

SUMMARY:
An observational study of patients with emerging or established severe cerebral vasospasm after subarachnoid haemorrhage, employing multimodal neuromonitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Critical care after subarachnoid haemorrhage
* Aneurysm secured by surgical clipping or endovascular procedure
* Suspected, emerging or established severe cerebral vasospasm

Exclusion Criteria:

* Anticipated survival less than five days, as determined by treating clinician
* Transcranial Doppler signal too weak
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for subarachnoid haemorrhage at the Intensive care unit at Karolinska University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Flow Velocity (MFV) | Up to 12 hours post intervention
  Increase or decrease of Mean Flow Velocity of the medial cerebral artery as determined by Transcranial Doppler.

SECONDARY OUTCOMES:
Duration of MFV change after Endoluminal Spasmolysis | Up to 12 hours
  Time until Mean Flow Velocity, as determined by Transcranial Doppler, returns to or surpasses baseline.

OTHER OUTCOMES:
Associations between Mean Flow Velocity and multimodal neurophysiologic measurement variables after endoluminal spasmolysis or induced hypertension. | Up to 12 hours
  Associations between Mean Flow Velocities, as determined by Transcranial Doppler, and other neurophysiologic measurement variables, such as pbtO2 (partial pressure brain tissue oxygenation), SbtO2 (brain tissue saturation), qEEG (quantitative EEG), microdialysis parameters, Prx (pressure reactivity index), as well as other physiologic output parameters such as cardiac output, (as determined by left ventricular output or effective pulmonary blood flow (EPBF)).
Associations between Mean Flow Velocity and neuroradiological outcome after induced hypertension or endoluminal spasmolysis. | Up to 12 hours
  Associations between Mean Flow Velocity, as determined by Transcranial Doppler, and neuroradiologic outcome parameters such as cerebral artery diameter, perfusion parameters, mean transit time (MTT), ischemic burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Observational, hypothesis-generating study.

DOCUMENTS (1):
  • Study Protocol (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT07305922/Prot_000.pdf